CLINICAL TRIAL: NCT05984199
Title: Phase 1/2 Study of Donor-Derived Anti-CD33 Chimeric Antigen Receptor Expressing T Cells (VCAR33) in Patients With Relapsed or Refractory Acute Myeloid Leukemia After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Donor-Derived Anti-CD33 CAR T Cell Therapy (VCAR33) in Patients With Relapsed or Refractory AML After Allogeneic Hematopoietic Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBP301
Record Dates: First submitted 2023-07-19; First posted 2023-08-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia; Acute Myeloid Leukemia; AML; Hematopoietic stem cell transplant; HCT; CD33; Allogeneic; CAR T; CAR-T; Chimeric Antigen Receptor T Cell; CAR T Cells; CAR-T Cells; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Morphologic Disease: Cohort 1 (Experimental): VCAR33 Dose Level 1
  Interventions: Biological: VCAR33
- Morphologic Disease: Cohort 2 (Experimental): VCAR33 Dose Level 2
  Interventions: Biological: VCAR33
- Morphologic Disease: Cohort 3 (Experimental): VCAR33 Dose Level 3
  Interventions: Biological: VCAR33
- MRD Positive: Cohort 1 (Experimental): VCAR33 Dose Level 1
  Interventions: Biological: VCAR33
- MRD Positive: Cohort 2 (Experimental): VCAR33 Dose Level 2
  Interventions: Biological: VCAR33
- MRD Positive: Cohort 3 (Experimental): VCAR33 Dose Level 3
  Interventions: Biological: VCAR33

INTERVENTIONS:
Biological: VCAR33 — Allogeneic Anti-CD33 Chimeric Antigen Receptor (CAR) T Cell therapy

SUMMARY:
This is a Phase 1/2, multicenter, open-label, first-in-human (FIH) study of donor-derived anti-CD33 Chimeric Antigen Receptor (CAR) T cell therapy (VCAR33) in patients with relapsed or refractory Acute Myeloid Leukemia (AML) after human leukocyte antigen (HLA)-matched allogeneic hematopoietic cell transplant (alloHCT).

DETAILED DESCRIPTION:
CD33 is a preferential target for AML CAR T cell therapy due to its surface expression on the majority (>80%) of AML blasts and due to the extensive prior clinical experience demonstrating safety and efficacy of targeting CD33 with Mylotarg (gemtuzumab ozogamicin). VCAR33 is being developed as a potential new treatment for patients with relapsed/refractory (R/R) AML after alloHCT. In this Phase 1/2 trial, the safety and efficacy of lentiviral-transduced CD33-directed CAR T cells (VCAR33) generated from the patient's prior allogeneic stem cell donor will be tested. It is hypothesized that CAR T cell production from healthy donors will not only eliminate delays in production due to lymphopenia but also reduce concerns for suboptimal T cell function from exposure to systemic immunosuppression or chemotherapeutic agents. Approximately 24 eligible patients with R/R AML after alloHCT will be enrolled in one of two separate arms based on disease burden (morphologic disease versus measurable residual disease (MRD ) positive). The maximum tolerated dose of VCAR33 will be determined using a 3+3 trial design within each arm. Dose escalation can only occur after a minimum of 3 patients have completed the dose-limiting toxicity (DLT) observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years
2. Patients must have CD33+ AML in relapse or refractory after alloHCT
3. Patients must be a recipient of an 8/8 (A, B, C, DRB1) HLA-matched related or unrelated donor alloHCT. Patients previously transplanted with VOR33 in the VBP101 study who have R/R AML may also be considered.
4. Disease status at the time of enrollment:

   1. Arm A/Morphologic disease: Defined as ≥ 5% blasts (bone marrow) post-HCT
   2. Arm B/MRD positive: < 5% blasts (bone marrow) with minimal residual disease of at least 0.1% CD33+ leukemia cells by flow cytometry
5. Performance status: ECOG 0 or 1
6. Patient must have adequate organ function as defined by:

   1. Cardiac: Left ventricular ejection fraction (LVEF) ≥ 45% or fractional shortening ≥ 28%
   2. Pulmonary: Baseline oxygen saturation > 92% on room air at rest
   3. Hepatic: Total bilirubin < 3x institutional upper limit of normal (ULN) (except in case of patients with documented Gilbert's disease < 5x ULN) and aspartate aminotransferase (AST/SGOT)/alanine aminotransferase (ALT/SGPT) < 5x institutional ULN
   4. Renal: Serum creatinine must be ≤ 1.2x institutional ULN or creatinine clearance ≥ 60 mL/min for patients with creatinine levels above institutional normal
7. Original alloHCT donor is available and willing to undergo apheresis

Exclusion Criteria:

1. Patients who have undergone more than one alloHCT
2. Patients who have undergone alloHCT with a mismatched unrelated donor, haploidentical donor, or with umbilical cord blood as the stem cell source
3. Patients who will be less than 100 days post-alloHCT at the time of VCAR33 infusion.
4. Patients with any history of Grade III or IV acute GVHD or severe chronic GVHD unless approved by the Sponsor Medical Monitor
5. Patients with evidence of ongoing active acute or chronic GVHD and are taking systemic immunosuppressive agents (> 10 mg daily of prednisone equivalent or other GVHD-directed treatment, including extracorporeal photopheresis). Patients with Grade 1 acute GVHD limited to the skin or mild chronic GVHD limited to the eyes, mouth, or skin controlled with only topical therapy are eligible.
6. Patients with active CNS disease. A lumbar puncture is not required to exclude CNS disease in the absence of clinical signs or symptoms suggesting CNS disease.
7. Patients with the following prior therapy:

   1. DLI within 28 days prior to enrollment
   2. Prior treatment with any CAR T cell therapy product
8. Patients with active or uncontrolled viral, bacterial, or fungal infection
9. Patients with a history of a human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection
10. Patients with a history of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, or breast) unless disease free for at least 3 years after the last definitive therapy
11. Female patients of childbearing potential who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Day 28

SECONDARY OUTCOMES:
Incidence of GVHD related to VCAR33 | Up to 24 months
Percentage of patients who achieve response | Up to 24 months
Overall survival post-VCAR33 infusion | Up to 24 months
Progression-free survival post-VCAR33 infusion | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute, Stanford, California
  - Miami Cancer Institute, Miami, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - The University of Kansas Cancer Center, Fairway, Kansas
  - National Institutes of Health, Clinical Center, Bethesda, Maryland
  - University of Michigan Health, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Mushtaq MU, DiPersio JF, Azzi J, Cooper BW, Koehne G, Koura D, Maakaron JE, Magenau JM, McClune B, Rimando JC, Shah NN, Suh HC, Beuka K, Sturrock J, Nikam MH, Berglund E, Hu J, Keschner Y, Etchin J, Lydeard JR, Vasquez MD, O'Donnell D, Mundelboim G, Thosar S, Canesin G, Xavier-Ferrucio J, Hyzy SL, Lloyd DM, Spink K, Hummel D, Lee-Sundlov MM, Scherer J, Lin MI, Whangbo JS, Muffly LS. A phase 1/2 study of donor-derived anti-CD33 CAR T-cell therapy (VCAR33) for relapsed/refractory AML after allogeneic HCT. Blood. 2026 Feb 4:blood.2025031053. doi: 10.1182/blood.2025031053. Online ahead of print. PMID 41636724